CLINICAL TRIAL: NCT04884828
Title: Trigger Asynchronies Induced by the Introduction of External Gas Into the Non-invasive Mechanical Ventilation Circuit: a Bench-to-bedside Study
Brief Title: Asynchronies in NIV With External Gas
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Cristina Lalmolda-Puyol, Respiratory therapist, Corporacion Parc Tauli
Other Study IDs: gasNIV
Record Dates: First submitted 2021-05-03; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Non-invasive Ventilation
Keywords: Non-invasive Ventilation; trigger asynchronies; autotriggering; bench study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one group: patients from the Pulmonology Service of the Corporació Sanitària Parc Taulí (Sabadell, Barcelona) who met the following criteria: over 18 years of age, hospital admission for acute chronic respiratory failure, home NIV (single-limb system with intentional leakage) users for more than 6 months with adequate compliance (greater than or equal to 5 hours/night). Patients with underlying psychiatric disease were excluded. The study was conducted during the patient's predischarge phase (the same day or the day before)
  Interventions: Device: external gas during NIV

INTERVENTIONS:
Device: external gas during NIV — The procedure was performed in the patient's room during his or her hospital stay to avoid additional visits for study participation. The patient was placed in the supine position, and the usual ventilator interface was placed in a single-limb system, along with the commercial ventilator to be studied. The ventilator model were evaluated at bedside in random order. The parameters of the ventilator were the same as those that the patients used at home (that is, unlike the bench study, the sensitivity of the trigger was not modified). A external polygraph was used to moritor the study, with the incorporation of thoracic and abdominal bands and parasternal electromyography, to better evaluate asynchronies, in addition to pulse oximetry control. The ventilation periods were 1 minute (without gas, gas, without gas). This sequence was performed twice in each group of established conditions.

SUMMARY:
NIV can be combined with other treatments that require to introduce gas into the circuit during the treatment. This external gas produces trigger asynchronies that worse depending on the model ventilator, trigger design and gas source. It is advisable to monitor NIV when these treatments are requiring in chronic NIV.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* hospital admission for acute chronic respiratory failure,
* home NIV (single-limb system with intentional leakage) users for more than 6 months with adequate compliance (greater than or equal to 5 hours/night).

Exclusion Criteria:

* Patients with underlying psychiatric disease were excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from the Pulmonology Service of the Corporació Sanitària Parc Taulí (Sabadell, Barcelona) who met the following criteria: over 18 years of age, hospital admission for acute chronic respiratory failure, home NIV (single-limb system with intentional leakage) users for more than 6 months with adequate compliance (greater than or equal to 5 hours/night). Patients with underlying psychiatric disease were excluded. The study was conducted during the patient's predischarge phase (the same day or the day before)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Asynchronies ( yes or no) | 1 day
  Presence of asynchronies identify by SOMNONIV´s algorithm during the gas treatment with NIV
Type of asynchronies | 1 day
  autotrigger or innefective effort identify by SOMNONIV´s group algorithm, during the gas treatment with NIV

SECONDARY OUTCOMES:
Type of asynchronies pre | 1 day
  autotrigger or innefectuve effort identify by SOMNONIV´s group pre gas during NIV treatment
Type of asynchronies post | 1 day
  autotrigger or innefective effort identify by SOMNONIV´s group algorithm, , post gas during NIV
Asynchronies ( yes or no) pre | 1 day
  Presence of asynchronies identify by SOMNONIV´s algorithm during pre-gas treatment with NIV
Asynchronies ( yes or no) post | 1 day
  Presence of asynchronies identify by SOMNONIV´s algorithm during the post gas treatment with NIV

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Lalmolda, RT PhD, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Cristina Lalmolda, Sabadell, Barcelona, Spain